CLINICAL TRIAL: NCT03239938
Title: Contemporary Pain Neuroscience Compared to Usual Care Evidence-based Physiotherapy Applied to Chronic Pain in Patients With Chronic Whiplash Associated Disorders: Can we Decrease Central Sensitization?
Brief Title: Modern Pain Neuroscience Applied to Chronic Pain in Patients With Chronic Whiplash Associated Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: University Hospital, Ghent (Other); University Ghent (Other); Research Foundation Flanders (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Iris Coppieters, dr. Iris Coppieters (principal investigator), Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G007217N
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Whiplash
Keywords: chronic whiplash associated disorders; central sensitization; electroencephalography; physiotherapy; chronic pain; functionality; quality of life; stress management; randomized controlled trial; modern neuroscience approach; pain neuroscience education; neck school; exercise therapy; pain cognitions
MeSH Terms: conditions — Whiplash Injuries; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The trial will randomize 120 patients with chronic WAD, aged between 18 and 65 years, to the experimental (modern neuroscience approach including 3 sessions of therapeutic pain neuroscience education followed by 15 sessions of dynamic and functional cognition-targeted exercise therapy and stress management techniques (n = 60)) or the control treatment (usual care physiotherapy: 3 sessions of neck school followed by 15 sessions of exercise therapy focusing on strength, flexibility, endurance, and ergonomic principles (n= 60)).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modern pain neuroscience approach (Experimental): Modern pain neuroscience approach
  Interventions: Behavioral: Modern pain neuroscience approach
- Usual care evidence-based physiotherapy (Active Comparator): Usual care physiotherapy
  Interventions: Behavioral: Usual care evidence-based physiotherapy

INTERVENTIONS:
Behavioral: Modern pain neuroscience approach — The modern pain neuroscience approach includes 3 sessions (1 group and 2 individual sessions) of therapeutic pain neuroscience education followed by 15 individual sessions of dynamic and functional cognition-targeted exercise therapy and stress management techniques. In addition, participants will be instructed to perform a daily set of home exercises. The exercises will be performed in a time-contingent way. The 18 sessions will be spread over a period of 16 weeks.
  Arms: Modern pain neuroscience approach
Behavioral: Usual care evidence-based physiotherapy — The usual care evidence-based physiotherapy includes 3 sessions (1 group and 2 individual sessions) of neck school followed by 15 individual sessions of graded and active exercise therapy focusing on strength, flexibility, endurance, and ergonomic principles. In addition, participants will be instructed to perform a daily set of home exercises. The exercises will be performed in a symptom-contingent way. The 18 sessions will be spread over a period of 16 weeks.
  Arms: Usual care evidence-based physiotherapy

SUMMARY:
Modern pain neuroscience has advanced our understanding of chronic whiplash associated disorders (WAD). Previous studies have shown the importance of central sensitization, characterized by hypersensitivity of the somatosensory system, in explaining poor treatment outcome. Therefore, and to address the need for a better treatment of chronic WAD, we recently proposed a modern neuroscience approach to chronic WAD. Such approach includes two specific parts: therapeutic pain neuroscience education followed by dynamic and functional cognition-targeted exercise therapy and stress management techniques.

The primary scientific objective of the study entails examining the effectiveness of a modern neuroscience approach versus usual care evidence-based physiotherapy for reducing dysfunctioning in patients with chronic WAD. The secondary scientific objective of the study entails examining the effectiveness of a modern neuroscience approach versus usual care evidence-based physiotherapy for reducing pain, central sensitization, psychosocial problems, and socio-economic burden in patients with chronic WAD. The trial will randomize 120 patients with chronic WAD, aged between 18 and 65 years, to the experimental (modern pain neuroscience approach including 3 sessions of therapeutic pain neuroscience education followed by 15 sessions of dynamic and functional cognition-targeted exercise therapy and stress management techniques (n = 60)) or the control treatment (usual care physiotherapy including 3 sessions of neck school followed by 15 sessions of graded and active exercise therapy focusing on strength, flexibility, endurance, and ergonomic principles (n= 60)). The primary outcome measure is self-reported functional status. Secondary outcome measures include pain, health-related quality of life, psychological correlates, measures of central sensitization, and socio-economic factors. In addition, quantitative scalp Electroencephalography (EEG) to measure various parameters of brain activation will be performed during a conditioned pain modulation paradigm. Baseline assessment of all outcome measures will be performed.

Follow-up assessments will be performed immediately after 16 weeks of therapy (all tests), and 6 months (all tests) and 12 months (only questionnaires) after finishing the therapeutic intervention.

To investigate these objectives, a multi-center triple-blind randomized, controlled trial with 1 year follow up will be performed.

DETAILED DESCRIPTION:
Modern pain neuroscience has advanced our understanding of chronic whiplash associated disorders (WAD). Previous studies have shown the importance of central sensitization, characterized by hypersensitivity of the somatosensory system, in explaining poor treatment outcome. Therefore, and to address the need for a better treatment of chronic WAD, we recently proposed a modern neuroscience approach to chronic WAD. Such approach includes two specific parts: 3 sessions of therapeutic pain neuroscience education followed by 15 sessions of dynamic and functional cognition-targeted exercise therapy and stress management techniques. The main principles of cognition-targeted are the following: All exercises should be performed in a time-contingent ("Perform this exercise 10 times, regardless of the pain") rather than in a symptom-contingent way ("Stop or adjust the exercise when it hurts"). Goal setting is essentially done together with the patient, focussing on functionality. The treating physical therapist should continuously assess and challenge the patients' cognitions and perceptions about the pain and the anticipated outcome of each exercise, to change maladaptive cognitions and perceptions into positive ones.

The primary scientific objective of the study entails examining the effectiveness of a modern pain neuroscience approach versus usual care evidence-based physiotherapy for reducing dysfunctioning in patients with chronic WAD. The secondary scientific objective of the study entails examining the effectiveness of a modern neuroscience approach versus usual care evidence-based physiotherapy for reducing pain, central sensitization, psychological problems, and socio-economic burden in patients with chronic WAD. The trial will randomize 120 patients with chronic WAD, aged between 18 and 65 years, to the experimental (modern pain neuroscience approach (n = 60)) or control treatment (usual care evidence-based physiotherapy: 3 sessions of neck school followed by 15 sessions of graded and active exercise therapy focusing on strength, flexibility, endurance, and ergonomic principles (n= 60)). The primary outcome measure is functional status. Secondary outcome measures include pain, health-related quality of life, psychological correlates, socio-economic factors, and measures of central sensitization, including electrical detection and electrical pain thresholds measured with a constant current electrical stimulator, endogenous pain facilitation (temporal summation of electrical pain), endogenous pain inhibition assessed by the conditioned pain modulation paradigm (electrical stimulation as test stimulus and the cold pressor test (immersion of one hand in cold water of 12°C) as conditioning stimulus). In addition, quantitative scalp Electroencephalography (EEG) to measure various parameters of brain activation will be performed during the conditioned pain modulation paradigm.

To comply with these scientific objectives, the 120 chronic WAD patients will be subjected to the baseline assessment of all outcome measures.

Follow-up assessments will be performed immediately after 16 weeks of therapy (all tests), and 6 months (all tests) and 12 months (only questionnaires) after finishing the therapeutic intervention.

To investigate these objectives, a muli-center triple-blind randomized, controlled trial with 1 year follow up will be performed.

Appropriate statistical analyses will be performed to evaluate and compare treatment effects. Statistical, as well as clinical significant differences will be defined and the effect size will be determined. Relations between functional status, pain, psychological correlates and central sensitization will be investigated. Furthermore, prediction of pain and functional status by central sensitization and psychological correlates will be performed in chronic WAD patients. Also, factors associated with clinically important changes in the outcome measures will be unraveled. In addition, factors associated with poor outcome following treatment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a whiplash trauma which is at least 3 months old and causes pain since at least 3 months, with pain experience with a mean pain frequency of 3 or more days per week, and with self-reported moderate to severe pain-related disability, established by a score of 15 or more of a maximum of 50 on the Neck Disability Index
* Patients classified as WAD II or WAD III on the modified Quebec Task Force Scale
* Native Dutch speaker
* Not starting new treatments or medication and continuing their usual care 6 weeks prior to and during study participation (to obtain a steady state)
* Refraining from non-opioid analgesics in the previous 48h of the assessments
* Refraining from caffeine, alcohol, and nicotine in the previous 24h of the assessments

Exclusion Criteria:

* Neuropathic pain
* Being pregnant or having given birth in the preceding year
* Chronic fatigue syndrome
* Fibromyalgia
* Cardiovascular disorders
* Epilepsy
* Endocrinological disorders
* Rheumatic disorders
* Psychiatric disorders
* History of neck surgery
* Loss of consciousness during/after the whiplash trauma
* Post-traumatic amnesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Self-reported functional status or disability | The change between the baseline assessment and the 6 months follow-up assessment (6 months after the end of the therapy)
  The Dutch version of the Neck Disability Index (questionnaire)

SECONDARY OUTCOMES:
Self-reported functional status or disability | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T3 follow-up assessment 12 months after the end of the therapy.
  The Dutch version of the Neck Disability Index (questionnaire)
Self-reported health-related quality of life | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy, T3 assessment 12 months after the end of the therapy.
  The Dutch version of the Short Form Health Survey-36 items (questionnaire)
Self-reported pain assessment | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy, T3 follow-up assessment 12 months after the end of the therapy.
  A 0-10 Numeric Rating Scale for pain (questionnaire). Patients fill out the Numeric Rating Scale (0 no pain - 10 worst pain imaginable) for their perceived neck pain.
Self-reported central sensitization symptoms | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy, T3 follow-up assessment 12 months after the end of the therapy.
  The Dutch version of the Central Sensitization Inventory (questionnaire)
Electrical detection and electrical pain thresholds with a constant current electrical stimulator (DS7A Digitimer) | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy
  Determination of the electrical detection and electrical pain threshold with the electrical stimulator will be performed at the sural nerve of the dominant leg and at the median nerve of the dominant arm.
Endogenous pain facilitation assessed by a temporal summation paradigm | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy
  Temporal summation of electrical pain will be assessed by delivering 20 electrical stimuli at the intensity of the electrical pain threshold.
Endogenous pain inhibition assessed by a conditioned pain modulation paradigm | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy
  Conditioned pain modulation will be tested with electrical stimulation as test stimulus and the cold pressor test (immersion the hand up to the wrist in cold water of 12°C) as conditioning stimulus.
Quantitative Electroencephalography (QEEG) (Sienna digital EEG, EMS Biomedical, Korneuburg, Austria) will be recorded from 32 Sn surface electrodes using an electrode cap (Headcap, Expertise in Medical Solutions Biomedical, Korneuburg, Austria). | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy
  During the condition pain modulation paradigm a QEEG will be administered to examine various brain activity parameters.
Self-reported psychological correlates: Pain catastrophizing | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy, T3 follow-up assessment 12 months after the end of the therapy.
  The Dutch version of the Pain Catastrophizing Scale (questionnaire)
Self-reported psychological correlates: Illness perceptions | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy, T3 follow-up assessment 12 months after the end of the therapy.
  The Dutch version of the illness perception questionnaire-revised (questionnaire)
Self-reported psychological correlates: Post-traumatic stress | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy, T3 follow-up assessment 12 months after the end of the therapy.
  The Dutch version of the Impact of Event Scale revised (questionnaire)
Self-reported psychological correlates: Pain-related fear and fear-avoidance behaviour | Baseline assessment, T1 follow-up assessment after 16 weeks of therapy, T2 follow-up assessment 6 months after the end of the therapy, T3 follow-up assessment 12 months after the end of the therapy.
  The Dutch version of the Pain anxiety symptoms scale (PASS-20) (questionnaire)
Socio-economic factors | Baseline assessment, T2 follow-up assessment 6 months after the end of the therapy, T3 follow-up assessment 12 months after the end of the therapy, 1 year before enrollment in the study
  Self-reported questionnaire and data including health-care expenditure from publicly funded healthcare organizations.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Coppieters, PhD, Study Director — Vrije Universiteit Brussel; Jo Nijs, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (3):
- Belgium (3):
  - Sint-jozefkliniek Campus Bornem (AZ Rivierenland), Bornem, Antwerpen
  - Ghent University, Ghent, Oost-Vlaanderen
  - Vrije Universiteit Brussel, Brussels

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michaleff ZA, Maher CG, Lin CW, Rebbeck T, Jull G, Latimer J, Connelly L, Sterling M. Comprehensive physiotherapy exercise programme or advice for chronic whiplash (PROMISE): a pragmatic randomised controlled trial. Lancet. 2014 Jul 12;384(9938):133-41. doi: 10.1016/S0140-6736(14)60457-8. Epub 2014 Apr 4. PMID 24703832
- [Background] Pinheiro ES, de Queiros FC, Montoya P, Santos CL, do Nascimento MA, Ito CH, Silva M, Nunes Santos DB, Benevides S, Miranda JG, Sa KN, Baptista AF. Electroencephalographic Patterns in Chronic Pain: A Systematic Review of the Literature. PLoS One. 2016 Feb 25;11(2):e0149085. doi: 10.1371/journal.pone.0149085. eCollection 2016. PMID 26914356
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Paul L. Evidence for central sensitization in chronic whiplash: a systematic literature review. Eur J Pain. 2013 Mar;17(3):299-312. doi: 10.1002/j.1532-2149.2012.00193.x. Epub 2012 Sep 25. PMID 23008191
- [Background] Sterling M, Kenardy J. Physical and psychological aspects of whiplash: Important considerations for primary care assessment. Man Ther. 2008 May;13(2):93-102. doi: 10.1016/j.math.2007.11.003. Epub 2008 Jan 24. PMID 18221907
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Truijen S, Craps J, Van den Keybus N, Paul L. Pain neurophysiology education improves cognitions, pain thresholds, and movement performance in people with chronic whiplash: a pilot study. J Rehabil Res Dev. 2011;48(1):43-58. doi: 10.1682/jrrd.2009.12.0206. PMID 21328162
- [Background] Nijs J, Ickmans K. Chronic whiplash-associated disorders: to exercise or not? Lancet. 2014 Jul 12;384(9938):109-11. doi: 10.1016/S0140-6736(14)60130-6. Epub 2014 Apr 4. No abstract available. PMID 24703833
- [Background] Dolphens M, Nijs J, Cagnie B, Meeus M, Roussel N, Kregel J, Malfliet A, Vanderstraeten G, Danneels L. Efficacy of a modern neuroscience approach versus usual care evidence-based physiotherapy on pain, disability and brain characteristics in chronic spinal pain patients: protocol of a randomized clinical trial. BMC Musculoskelet Disord. 2014 May 8;15:149. doi: 10.1186/1471-2474-15-149. PMID 24885889
- [Background] Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. Aust J Physiother. 2002;48(4):297-302. doi: 10.1016/s0004-9514(14)60169-0. PMID 12443524
- [Background] Meeus M, Nijs J, Hamers V, Ickmans K, Oosterwijck JV. The efficacy of patient education in whiplash associated disorders: a systematic review. Pain Physician. 2012 Sep-Oct;15(5):351-61. PMID 22996847
- [Background] Nijs J, Lluch Girbes E, Lundberg M, Malfliet A, Sterling M. Exercise therapy for chronic musculoskeletal pain: Innovation by altering pain memories. Man Ther. 2015 Feb;20(1):216-20. doi: 10.1016/j.math.2014.07.004. Epub 2014 Jul 18. PMID 25090974
- [Background] Southerst D, Nordin MC, Cote P, Shearer HM, Varatharajan S, Yu H, Wong JJ, Sutton DA, Randhawa KA, van der Velde GM, Mior SA, Carroll LJ, Jacobs CL, Taylor-Vaisey AL. Is exercise effective for the management of neck pain and associated disorders or whiplash-associated disorders? A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Spine J. 2016 Dec;16(12):1503-1523. doi: 10.1016/j.spinee.2014.02.014. Epub 2014 Feb 15. PMID 24534390
- [Background] Nijs J, Meeus M, Cagnie B, Roussel NA, Dolphens M, Van Oosterwijck J, Danneels L. A modern neuroscience approach to chronic spinal pain: combining pain neuroscience education with cognition-targeted motor control training. Phys Ther. 2014 May;94(5):730-8. doi: 10.2522/ptj.20130258. Epub 2014 Jan 30. PMID 24481595
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Derived] Malfliet A, Lenoir D, Murillo C, Huysmans E, Cagnie B, Meeus M, Willaert W, Ickmans K, Danneels L, Bontinck J, Nijs J, Coppieters I. Pain Science Education, Stress Management, and Cognition-Targeted Exercise Therapy in Chronic Whiplash Disorders: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2526674. doi: 10.1001/jamanetworkopen.2025.26674. PMID 40794407